CLINICAL TRIAL: NCT04603196
Title: Prevalence and Impact of Obstructive Sleep Apnea in Multiple Sclerosis
Acronym: SOMNUS
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Jacob Sloane, Assistant Professor of Neurology, Beth Israel Deaconess Medical Center
Other Study IDs: 2019P000494
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Obstructive Sleep Apnea
MeSH Terms: conditions — Multiple Sclerosis; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with Multiple Sclerosis with obstructive sleep apnea: Patients with Multiple Sclerosis with obstructive sleep apnea
- Patients with MS without obstructive sleep apnea: Patients with MS without obstructive sleep apnea

SUMMARY:
This study will evaluate the influence of sleep apnea on clinical and radiological features of MS. Sleep apnea is associated with hypoxemia during sleep, which is likely detrimental to MS. Clinical data (MRI, lab results, medical history, labs, and sleep studies) of MS patients will be collected and analyzed. This will be done to study correlations between MRI, clinical data, lab studies and sleep studies. There is specific interest in the type of sleep apnea associated with MS, and whether MRI or clinical metrics of MS severity correlate with presence or absence of sleep apnea.

DETAILED DESCRIPTION:
BACKGROUND Multiple sclerosis (MS) is an inflammatory demyelinating neurologic disease associated with significant disability. Many pathological mechanisms are believed to drive MS, including inflammation. However, the mechanism behind progression, the major driver of disability in MS, is thought to be distinctly different. With progression, neurodegeneration and loss of neurons/axons appears to be primarily responsible. A theory of "virtual hypoxia" has been theorized, in that inflammation and demyelination cause neurons and axons to work harder, utilizing more energy. The overuse of neuron/axon energy makes it more likely that there are periods of low/absent energy availability, which drives neuron/axon degeneration and progression in MS.

It is well known that MS is associated with sleep apnea. Obstructive sleep apnea (OSA) prevalence in MS patients is approximately 58%. Sleep apnea is a disorder where lower blood oxygenation occurs during sleep. Since it is probable that low blood oxygenation would contribute to neuron/axon injury, it is possible MS patients with sleep apnea have worse neurological outcomes (clinically and radiographically).

It is possible that testing can show an effect on neuron/axon injury as well as inflammation. In addition to MRI changes that correlate with these changes, there are blood markers of neurodegeneration and inflammation including neurofilament-light (NFL) and glial fibrillary acidic protein (GFAP), now available for blood testing commercially. Elevations in such markers may be associated with sleep apnea.

This study will enable a first approximation of the prevalence of sleep apnea in MS as well as associated features of the comorbidity.

Patients will undergo a Home Sleep Test study using an at home polysomnagraphy device to help determine an accurate prevalence rate of sleep apnea in the MS population. Patients will also answer questionnaires to gain qualitative data on fatigue, sleepiness, sleep quality, restless leg syndrome risk, pain, sleep apnea risk, depression, and anxiety. Lastly, blood samples will be collected to study markers of neurodegeneration and inflammation.

B3. DESCRIPTION OF RESEARCH PROTOCOL A. Study Design - Overview, Methods, Procedures

Study Participants Subjects with a confirmed diagnosis of multiple sclerosis will be the inclusion criteria for this study. As patients come to clinic for their routine clinical care visits, MS patients will be recruited. During these visits patients will be identified through their medical records those who are pre- treatment for OSA with CPAP (Continuous Positive Airway Pressure) machine and those who are currently on this therapy.

The plan is to identify approximately 400 people will take part in this study at Beth Israel Deaconess Medical Center. Approximately 200 people each will take part in this study at UMass Medical Center MS Center and at Lahey MS Center. A total of 800 people will take part in this study at all study sites.

Study Procedures

Medical Record Review Retrospective data from the patient's medical record will be collected including date of birth and demographic data. Past medical history including medical conditions, surgical history, family history, social history, medications, allergies, as well as the results from prior neurological exams, diagnostic tests, MRIs, previous lab work, and genetic testing will also be collected.

Clinical Information Collection Clinical information from routine clinical care visits will be collected including medical history, surgical history, family history, social history, medications, and allergies. Study sites will also collect other information including vital signs, results from diagnostic tests including lab work and MRIs, neurological exams, neurological and physical functioning assessments on their level of disability, cognitive functioning, hand eye coordination, vision, and walking ability,

Questionnaires Questionnaires will be used to assess sleep quality and habits, urinary habits, risk of sleep apnea, fatigue levels, insomnia levels, risk of restless leg syndrome, depression, anxiety, and pain levels. They will take approximately 60 minutes to complete.

Body Measurements. Neck size, height and weight will be measured and BMI will be calculated

Blood Sample Collection Blood will be taken at their screening clinical care visit, at month 6, and month 12. The number of samples and the amount of blood collected will vary at each visit but will not exceed 5ml per visit. Markers of neurodegeneration and inflammation including neurofilament-light (NFL) and glial fibrillary acidic protein (GFAP) will be measured.

Home Sleep Test Subjects will undergo a home sleep test to assess for sleep apnea. The Home Sleep Test (HST) is a device that has an oximeter, a string that goes around the chest to record breaths. The HST device also has a lightweight tube which on one end splits into two prongs which are placed in the nostrils for measuring air movement. Within one month of their screening visit, subjects will wear the wrist oximeter and the HST device overnight while subjects sleep and remove them upon waking in the morning. Subjects will only do this once. Subjects then either return the device to the clinic in person or mail the device back using pre-addressed and pre-paid packaging within one week of completing the test.

Schedule of Study Activities

Screening:

* Informed consent
* Confirming MS diagnosis
* Height, weight, neck size measurement
* Questionnaires: Sleep History (NDSQ), STOP-BANG, Berlin, Modified Fatigue Impact Scale (MFIS), Fatigue Severity Scale (FSS), Epworth Sleepiness Scale (ESS), Insomnia Severity Index (ISI), Pittsburgh Sleep Quality Index (PSQI), Restless Legs Syndrome-Diagnostic Index (RLS-DI), Pain Scale (NRS), and Hospital Anxiety and Depression Scale (HADS)
* Blood draw

Within 1 month of screening • Home Sleep Study

Month 6:

* Questionnaires: STOP-BANG, Berlin, MFIS, FSS, ESS, ISI, PSQI, RLS-DI, and HADS
* Blood draw

Month 12

* Questionnaires: STOP-BANG, Berlin, MFIS, FSS, ESS, ISI, PSQI, RLS-DI, and HADS
* Blood draw

Data Analysis

• Data will be analyzed continually over the course of this study. Once HST data is collected the investigators will determine sleep apnea prevalence and severity. HST data will be correlated with questionnaire findings and clinical metrics of MS disease activity/disability.

Research Activities as Coordinating Site:

The coordinating site will train the other involved sites in accordance with the protocol. All sites will have a copy of our IRB approved protocol. BIDMC study site will communicate with the other sites on an as needed basis regarding updates to the protocol or any other changes to the study. Any retraining will be performed if requested. The coordinating site will provide questionnaires, checklists, and materials related to completion of the proposed work. The coordinating site will disseminate funds as required from any grant associated with this work.

The coordinating site will be in charge of collecting and storing all data for the proposed study. This data includes clinical and demographic data as well as laboratory and radiological data. The coordinating site will record any deviations and adverse events related to the protocol. The principle investigator will oversee all unanticipated problems, adverse events, noncompliance, and new information about the study will be report them to the other sites immediately.

B. Statistical Considerations

1. Sample Size Justification: All MS patients from BIDMC, UMASS, and Lahey Hospital systems are eligible for this study. The sample size will be 400 patients from Beth Israel Deaconness Medical Center, 200 from Lahey Clinic, and 200 from UMASS for 800 patients total.
2. Data Analysis: All data will be collected and stored using Microsoft Excel on a secure computer. Data analysis will be conducted by utilizing Harvard Catalyst biostatistician services. Statistical analyses used will be up to the discretion of the biostatistician and team.

C. Subject Selection Patients with MS will be identified via BIDM, Lahey, or UMASS electronic medical records and also to distinguish those who are either on CPAP therapy or not.

B4. POSSIBLE BENEFITS There is no direct benefit to the patient from being in this study. However, patients' participation may help others in the future as a result of knowledge gained from this database.

B5. POSSIBLE RISKS AND ANALYSIS OF RISK/BENEFIT RATIO There are minimal risks associated with this medical record review, which include a breach of confidentiality. The risk that someone other than the patient's physician and the MS treatment team will be able to link the patient's information to the study with the patient's name is minimal. Information will be kept in a secure, password-protected computer within the MS team's research drive.

Some of the questions asked as part of the study, may make the patient feel uncomfortable. They may refuse to answer any of the questions. Although not ideal for purposes of this study, refusing to answer questions/questionnaires is permissible.

HST devices are used as a diagnostic tool routinely in clinical practice for sleep apnea and are FDA approved for this indication. Complications are rare and not high-risk. The most common side effect is skin irritation caused by the adhesive used to attach test sensors to the skin.

Risk of blood draw may include discomfort, bruising, and very rarely infection at the site where the needle enters the skin. Patients may also possibly experience dizziness, nausea, or fainting during blood collection

RECRUITMENT Subjects will be identified via medical record review. Any subject data included in the study will be a result of the subject matching the inclusion criteria.

Consent

Written Consent The PI on this study has requested a HIPPA Waiver of Authorization due to the fact that this is a retrospective medical record review. An informed consent will be signed for the HST device substudy.

Verbal Consent Prior to any data collection under this protocol for patients restricted to telemedicine visits due to COVID-19, a verbal consent will be obtained using a verbal consent script. An information sheet will be sent to the patient by email or by mail. Written consent can be obtained if/when subjects come to the medical center for in person visits.

Subject Protection No subjects in this study will be vulnerable to coercion or undue influence because this is a retrospective medical record review. However, since this study does involve the use of PHI, every effort will be maintained to de-identify PHI to maintain confidentiality. In addition, each subject will be given a unique identifier (i.e. 001) and the codebreaker will be located in a secure, locked office

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Over age 18
* Confirmed diagnosis of multiple sclerosis

Exclusion Criteria:

* cannot provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a confirmed diagnosis of multiple sclerosis will be the inclusion criteria for this study. As patients come to clinic for their routine clinical care visits, the investigators will identify presence of MS.
  The investigators will identify approximately 400 people will take part in this study at Beth Israel Deaconess Medical Center. Approximately 200 people each will take part in this study at UMass Medical Center MS Center and at Lahey MS Center. A total of 800 people will take part in this study at all study sites.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2030-06-20 (Estimated)

PRIMARY OUTCOMES:
Home Sleep Study Data | 1 year
  Home Sleep Study Data

SECONDARY OUTCOMES:
Questionnaire data | 1 year
  sleep quality, quality of life, depression and anxiety scales

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States